CLINICAL TRIAL: NCT06087081
Title: Effects of Mills Manipulation With and Without Mulligan Pain Release Phenomena on Pain, Hand Grip Strength and Function in Patients With Lateral Epicondylitis
Brief Title: Mills Manipulation and Mulligan PRP Affect Pain, Grip Strength and Function on Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0144
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral Epicondylitis; Elbow; Pain; Tennis Elbow; Mills Manipulation; Mulligan; Pain Release Phenomena; Hand Grip Strength; Elbow Function; NPRS; PRTEE; Hand Held Dynamometer
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Baseline treatment along with Mill's manipulation
  Interventions: Other: Baseline Treatment along with Mill's manipulation
- Group B (Experimental): Baseline Treatment along with Mill's manipulation and Mulligan's pain relief phenomena
  Interventions: Other: Baseline Treatment along with Mill's manipulation and Mulligan's pain relief phenomena

INTERVENTIONS:
Other: Baseline Treatment along with Mill's manipulation — Position the patient on a chair with a backrest and stand behind the patient. Support the patient's arm under the crook of the elbow with the shoulder joint abducted to 90° and medially rotated. The forearm will automatically fall into pronation. Place the thumb of your other hand in the web space between the patient's thumb and index finger and fully flex the patient's wrist and pronate the forearm. Move the hand supporting the crook of the elbow on to the posterior surface of the elbow joint and, while maintaining full Wrist flexion and pronation, extend the patient's elbow until you feel that all the slack Has been taken up in the tendon. Step sideways to stand behind the patient's head, Taking Care to prevent the patient from leaning away either forwards or sideways, which would reduce the tension on the tendon.
  Each exercise will be done 10 times for 5 sets each with a rest interval of 10 seconds in between each set for a period of 4 weeks
  Arms: Group A
Other: Baseline Treatment along with Mill's manipulation and Mulligan's pain relief phenomena — In addition to Group A mentioned protocols Pain release phenomenon (PRP) was delivered as well. The Pain Release Phenomenon Technique (PRPS) is a technique pioneered by Brian Mulligan for management of Pain. There are different types of Pain release Phenomenon as follows:
  1. Stretch PRP: affected muscle is eccentrically contracted.
  2. Contraction PRP: affected muscle is concentrically contracted.
  3. Compression PRP: affected joint surfaces are compressed together.
  4. Distraction PRP: affected joint surfaces are distracted away from each other. The types of PRP are performed along with pertained duration of hold time by the therapist. And always painful PRP technique is chosen for the treatment. In the present study stretch PRP technique was used which provoked pain stimuli and was maintained for 15-20 seconds. Each exercise will be done 10 times for 5 sets each with a rest interval of 10 seconds in between each set for a period of 4 weeks
  Arms: Group B

SUMMARY:
The aim of this study is to find the comparative effects of mills manipulation with or without Mulligan pain release phenomena on the pain, grip strength, and function in patients with Lateral Epicondylitis. The results of this study will provide clinicians with valuable insights into the most effective treatment approach for lateral epicondylitis, enabling them to stay up-to-date with the latest practice methods and optimize patient care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with lateral epicondylitis with positive Cozen test
* NPRS >3
* Both male and female patients
* Sub-acute lateral epicondylitis >4weeks-<3 months
* Subjects with age range 20-40 year

Exclusion Criteria:

* Acute lateral epicondylitis
* Subjects with elbow and around elbow fracture
* Subjects with ligament injury around elbow joint
* Any neurological conditions
* Any open wounds around the area of elbow
* Hyper-sensitive skin, skin allergies, diagnosed subjects with malignancy, diagnosed subjects skin diseases, diagnosed subjects with systemic illness
* Traumatic injury to the elbow joint

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rate Scale | 4th Week
  The NPRS for pain is a unidirectional measure of pain intensity in adults similar to the pain Visual Analogue Scale(VAS), the NPRS is anchored by terms describing pain severity extremes. The common format is a horizontal bar or line with 11-items (0-10). 0 on NPRS indicates no pain, 5 indicates moderate pain and 10 indicates worst possible pain. NPRS is easy to administer and takes less than 1minute. The NPRS can be administered verbally (on telephone) or graphically for self- completion. Reliability: high test-retest reliability (r=0.96). Validity: (0.86-0.95).
Hand Held Dynamometer | 4th Week
  The maximal grip strength of the affected arm was assessed using a grip-strength dynamometer. Patients were asked to grip the dynamometer as hard as possible 3 times at 10 s rest interval. Grip force should be applied smoothly without rapid jerking motion. Patient must be seated with 90 degrees of elbow flexion, shoulder adduction, slight extension in the wrist, and the forearm in the neutral position. The highest grip-strength number was registered. Reliability: high test-retest reliability(r=0.9864)
Patient-Rated Tennis Elbow Evaluation | 4th Week
  Functional Disability was measured by PRTEE, a 15-item questionnaire designed to measure forearm pain and disability in patients with Lateral Epicondylitis. Patients have to rate their levels of tennis elbow pain and disability from 0 to 10 and consists of 2 sub-scales. There is a pain sub-scale with 5 items (0 = no pain, 50 = worst pain) and Functional sub-scale consists of Specific activities with 6 items (0 = no hinder, 60 =unable to do) and Usual activities with 4 items (0 = no difficulty, 10 = unable to do). The PRTEE was found to be a reliable, reproducible and sensitive instrument for the assessment of pain and disability in chronic lateral epicondylitis subjects (Cronbach's alpha is 0.98).

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar, MS, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital Trust, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker CL Jr, Murphy KP, Gottlob CA, Curd DT. Arthroscopic classification and treatment of lateral epicondylitis: two-year clinical results. J Shoulder Elbow Surg. 2000 Nov-Dec;9(6):475-82. doi: 10.1067/mse.2000.108533. PMID 11155299
- [Background] Armstrong TJ, Buckle P, Fine LJ, Hagberg M, Jonsson B, Kilbom A, Kuorinka IA, Silverstein BA, Sjogaard G, Viikari-Juntura ER. A conceptual model for work-related neck and upper-limb musculoskeletal disorders. Scand J Work Environ Health. 1993 Apr;19(2):73-84. doi: 10.5271/sjweh.1494. PMID 8316782
- [Background] Ahmad Z, Siddiqui N, Malik SS, Abdus-Samee M, Tytherleigh-Strong G, Rushton N. Lateral epicondylitis: a review of pathology and management. Bone Joint J. 2013 Sep;95-B(9):1158-64. doi: 10.1302/0301-620X.95B9.29285. PMID 23997125
- [Background] Bretschneider SF, Los FS, Eygendaal D, Kuijer PPFM, van der Molen HF. Work-relatedness of lateral epicondylitis: Systematic review including meta-analysis and GRADE work-relatedness of lateral epicondylitis. Am J Ind Med. 2022 Jan;65(1):41-50. doi: 10.1002/ajim.23303. Epub 2021 Oct 21. PMID 34674287
- [Background] Aldajah S, Alashram AR, Annino G, Romagnoli C, Padua E. Analgesic Effect of Extracorporeal Shock-Wave Therapy in Individuals with Lateral Epicondylitis: A Randomized Controlled Trial. J Funct Morphol Kinesiol. 2022 Mar 18;7(1):29. doi: 10.3390/jfmk7010029. PMID 35323612
- [Background] Fahmy FS, ElAttar M, Salem HF. Hand-Grip Strength and Return to Heavy Manual Work at a Mean 5-Year Follow-up After Arthroscopic Release of Recalcitrant Lateral Epicondylitis. Orthop J Sports Med. 2022 Feb 24;10(2):23259671221078586. doi: 10.1177/23259671221078586. eCollection 2022 Feb. PMID 35252465
- [Background] 8. Chintamani R. Effect of Mulligan's Pain Release Phenomenon on Ted in Subjects with Subacute Lateral Epicondylitis. Journal of Complementary and Alternative Medical Research. 2021;16(4):59-70.
- [Background] 1. Runge F. Zur genese und behandlung des schreibekrampfes. Berl Klin Wochenschr. 1873;10(1):245-8.
- [Background] 9. Sahu RK. A Comparative Study of Effectiveness of Mulligan's Mobilisation with Movement and Cyriax Deep Transverse Friction along with Mill's Manipulation in Individuals with Chronic Lateral Epicondylitis. 2020.
- [Background] 10. Memon AG, Latif FA, Sanaullah M, Hussain MI, Irum S, Rehman FU. Prevalence of lateral epicondylitis among restaurant chefs with low level of serum Vitamin D. Rawal Medical Journal. 2023;48(2):422-.
- [Background] 11. Zami MDZ, Pristianto A, Nasrullah N. The Effectiveness of Mulligan Mobilization With Movement (MWM) in Lateral Epicondylitis: a Critical Review. FISIO MU: Physiotherapy Evidences. 2023;4(1).
- [Background] 12. Rahman H, Chaturvedi PA, Apparao P, Srithulasi PR. Effectiveness of mulligan mobilisation with movement compared to supervised exercise program in subjects with lateral epicondylitis. Int J Physiotherapy Res. 2016;4(2):1394-400.